CLINICAL TRIAL: NCT02000427
Title: A Phase 2 Single Arm, Multicenter Trial to Evaluate the Efficacy of the BiTE Antibody Blinatumomab in Adult Subjects With Relapsed/Refractory Philadelphia Positive B-precursor Acute Lymphoblastic Leukemia (Alcantara Study)
Brief Title: Blinatumomab in Adults With Relapsed/Refractory Philadelphia Positive B-precursor Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120216; 2006-006520-19 (EudraCT Number)
Record Dates: First submitted 2013-11-15; First posted 2013-12-04 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Relapsed/Refractory Philadelphia Positive B-precursor ALL
Keywords: Relapsed; Refractory; Philadelphia Positive; B-precursor; Acute Lymphoblastic Leukemia; ALL; Blinatumomab; Leukemia;
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Participants will receive blinatumomab by continuous intravenous (CIVI) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for 2 cycles. Participants who achieve a complete remission or complete remission with partial or incomplete hematologic recovery within 2 induction cycles of treatment could receive up to 3 additional consolidation cycles of blinatumomab.
  The initial dose will be 9 μg/day for the first 7 days of treatment, increased to 28 μg/day starting on day 8 for all subsequent cycles of treatment.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is administered as a continuous intravenous infusion (CIV). A single cycle of blinatumomab treatment is 6 weeks in duration, which includes 4 weeks of blinatumomab followed by a 2-week treatment-free interval.
  Other Names: Blincyto®; AMG 103

SUMMARY:
The primary objective is to evaluate the rate of complete remission/complete remission with partial hematological recovery (CRh*) in adults with relapsed/refractory Philadelphia chromosome positive (Ph+) B-precursor acute lymphoblastic leukemia (ALL) who receive blinatumomab.

DETAILED DESCRIPTION:
This is a single-arm Simon II stage design, multicenter study consisting of a screening period, an induction treatment period (2 cycles of blinatumomab), a consolidation treatment period (up to 3 additional cycles of blinatumomab for applicable participants), and a safety follow-up visit 30 days after treatment. Following the safety follow-up visit, participants will be followed for response duration and survival every 3 months for 18 months or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Patients with Ph+ B-precursor ALL, with any of the following:

  * Relapsed or refractory to at least one second generation tyrosine kinase inhibitor (TKI) (dasatinib, nilotinib, bosutinib, ponatinib)
  * OR intolerant to second generation TKI and intolerant or refractory to imatinib mesylate
* Greater than 5% blasts in bone marrow
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Age ≥ 18 years of age, at the time of informed consent.
* Subject has provided informed consent or subject's legally acceptable representative has provided informed consent when the subject has any kind of condition that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent.

Exclusion Criteria

* History of malignancy other than ALL within 5 years prior to start of protocol-required therapy, except for adequately treated selected cancers without evidence of disease
* History or presence of clinically relevant central nervous system (CNS) pathology as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis
* Active ALL in the CNS or testes
* Isolated extramedullary disease
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Allogeneic hematopoietic stem cell transplantation (HSCT) within 12 weeks before blinatumomab treatment
* Active acute or extensive chronic graft-versus-host disease (GvHD) which included the administration of immunosuppressive agents to prevent or treat GvHD within 2 weeks before blinatumomab treatment
* immediately previous cancer chemotherapy, radiotherapy, or immunotherapy; and eligibility for allogeneic HSCT at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (8):
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Atlanta, Georgia
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Houston, Texas
- France (3):
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (4):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Würzburg
- Italy (5):
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Roma
  - Research Site, Venezia
  - Research Site, Verona
- United Kingdom (2):
  - Research Site, London
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinelli G, Boissel N, Chevallier P, Ottmann O, Gokbuget N, Topp MS, Fielding AK, Rambaldi A, Ritchie EK, Papayannidis C, Sterling LR, Benjamin J, Stein A. Complete Hematologic and Molecular Response in Adult Patients With Relapsed/Refractory Philadelphia Chromosome-Positive B-Precursor Acute Lymphoblastic Leukemia Following Treatment With Blinatumomab: Results From a Phase II, Single-Arm, Multicenter Study. J Clin Oncol. 2017 Jun 1;35(16):1795-1802. doi: 10.1200/JCO.2016.69.3531. Epub 2017 Mar 29. PMID 28355115
- [Background] Kuchimanchi M, Zhu M, Clements JD, Doshi S. Exposure-response analysis of blinatumomab in patients with relapsed/refractory acute lymphoblastic leukaemia and comparison with standard of care chemotherapy. Br J Clin Pharmacol. 2019 Apr;85(4):807-817. doi: 10.1111/bcp.13864. Epub 2019 Feb 18. PMID 30645768
- [Background] Kantarjian HM, Zugmaier G, Bruggemann M, Wood BL, Horst HA, Zeng Y, Martinelli G. Impact of Blinatumomab Treatment on Bone Marrow Function in Patients with Relapsed/Refractory B-Cell Precursor Acute Lymphoblastic Leukemia. Cancers (Basel). 2021 Nov 9;13(22):5607. doi: 10.3390/cancers13225607. PMID 34830762
- [Background] Clements JD, Zhu M, Kuchimanchi M, Terminello B, Doshi S. Population Pharmacokinetics of Blinatumomab in Pediatric and Adult Patients with Hematological Malignancies. Clin Pharmacokinet. 2020 Apr;59(4):463-474. doi: 10.1007/s40262-019-00823-8. PMID 31679130
- [Background] Martinelli G, Boissel N, Chevallier P, Ottmann O, Gokbuget N, Rambaldi A, Ritchie EK, Papayannidis C, Tuglus CA, Morris JD, Stein A. Long-term follow-up of blinatumomab in patients with relapsed/refractory Philadelphia chromosome-positive B-cell precursor acute lymphoblastic leukaemia: Final analysis of ALCANTARA study. Eur J Cancer. 2021 Mar;146:107-114. doi: 10.1016/j.ejca.2020.12.022. Epub 2021 Feb 13. PMID 33588145
- [Background] Topp MS, Stein AS, Gokbuget N, Horst HA, Boissel N, Martinelli G, Kantarjian H, Bruggemann M, Chen Y, Zugmaier G. Blinatumomab as first salvage versus second or later salvage in adults with relapsed/refractory B-cell precursor acute lymphoblastic leukemia: Results of a pooled analysis. Cancer Med. 2021 Apr;10(8):2601-2610. doi: 10.1002/cam4.3731. Epub 2021 Mar 18. PMID 33734596
- [Background] Horst HA, Zugmaier G, Martinelli G, Mergen N, Velasco K, Zaman F, Kantarjian H. CD19-negative relapse in adult patients with relapsed/refractory B-cell precursor acute lymphoblastic leukemia following treatment with blinatumomab-a post hoc analysis. Am J Hematol. 2023 Aug;98(8):E222-E225. doi: 10.1002/ajh.26988. Epub 2023 Jun 22. No abstract available. PMID 37345570
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 centers in 4 European countries and the United States: 3 centers in France, 3 in Germany, 5 in Italy, 1 in the United Kingdom, and 7 in the United States.
  The first participant enrolled on 03 January 2014 and the last participant enrolled on 12 January 2015.
Pre-assignment Details: Results are reported as of the data cut-off date of 20 May 2015.
Groups:
- Blinatumomab: Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for 2 cycles. Participants who achieved a complete remission or complete remission with partial or incomplete hematologic recovery within 2 induction cycles of treatment could receive up to 3 additional consolidation cycles of blinatumomab.
  The initial dose was 9 μg/day for the first 7 days of treatment, increased to 28 μg/day starting on day 8 and for all subsequent cycles of treatment.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 45
Completed | 23 (Indicates participants ongoing in study as of the data cut-off date of 20 May 2015.)
Not Completed | 22
Not completed — Death | 22

BASELINE CHARACTERISTICS:
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.0)
Age, Customized [Number; unit: participants]
  18 to < 35 years | 5
  35 to < 55 years | 17
  55 to < 65 years | 11
  ≥ 65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39
  Asian | 1
  Black (or African American) | 3
  Other | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 2
  Not Hispanic/Latino | 43
Prior Tyrosine Kinase Inhibitor (TKI) Treatment [Number; unit: participants]
  1 TKI | 7
  2 TKIs | 21
  3 TKIs | 13
  4 TKIs | 4
Number of Prior Relapses [Number; unit: participants]
  No relapses | 3
  1 relapse | 25
  2 relapses | 13
  ≥ 3 relapses | 4
Number of Prior Salvage Regimens [Number; unit: participants]
  0 regimens | 14
  1 regimen | 12
  2 regimens | 11
  ≥ 3 regimens | 8
Prior Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) [Number; unit: participants]
  Yes | 20
  No | 25
Time From Initial Diagnosis [Mean (Standard Deviation); unit: months] | 27.3 (26.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission/Complete Remission With Partial Hematological Recovery (CR/CRh*) During the First Two Treatment Cycles
Description: Participants were evaluated for efficacy at the end of each treatment cycle via a central bone marrow aspiration and local peripheral blood counts.
  Complete remission was defined as meeting all 3 of the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease
  * full recovery of peripheral blood counts: platelets > 100,000/μl, and absolute neutrophil count (ANC) > 1000/μl.
  Complete remission with partial hematological recovery (CRh*) was defined as meeting all 3 of the following criteria:
  * less than or equal to 5% blasts in the bone marrow
  * no evidence of disease
  * partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl.
  Participants without a post-baseline disease assessment were considered non-responders.
Time Frame: Approximately 12 weeks, as of the data cut-off date of 20 May 2015
Population: All participants who received an infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
percentage of participants | 35.6 [21.9 to 51.2]

2. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Remission During the First 2 Cycles of Treatment
Description: Bone marrow samples were evaluated for MRD remission by a central laboratory using bcr-abl fusion gene reverse transcription polymerase chain reaction (RT-PCR).
  An MRD response was defined as MRD < 10^-4 measured by PCR. Participants with no post-baseline MRD assessment were considered non-responders.
Time Frame: Approximately 12 weeks
Population: All participants who received an infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
percentage of participants | 40.0 [25.7 to 55.7]

3. Secondary Outcome: Duration of CR or CRh* Response
Description: Duration of response was measured for participants in remission (CR/CRh*), and was measured from the time the participant first achieved remission until first documented relapse or death from disease progression. Participants without a documented relapse (hematological or extramedullary) and who did not die were censored at the time of the last bone marrow assessment or the last survival follow-up visit to confirm remission. Participants who died without having reported hematological relapse or without showing any clinical sign of disease progression were censored on their date of death.
Time Frame: Up to the data cut-off date of 20 May 2015; median observation time was 7.0 months
Population: Participants who received an infusion of blinatumomab and with a CR or CRh* response during the first 2 treatment cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 16
months | 6.7 [4.5 to NA] — Could not be estimated due to the low number of events at the time of analysis

4. Secondary Outcome: Percentage of Participants With Complete Remission (CR) During the First Two Treatment Cycles
Description: Participants were evaluated for efficacy at the end of each treatment cycle via a central bone marrow aspiration and local peripheral blood counts.
  Complete remission was defined as meeting all 3 of the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease;
  * full recovery of peripheral blood counts: platelets > 100,000/μl, and absolute neutrophil count (ANC) > 1000/μl.
  Participants without a post-baseline disease assessment were considered non-responders.
Time Frame: Approximately 12 weeks, as of the data cut-off date of 20 May 2015
Population: All participants who received an infusion of blinatumomab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
percentage of participants | 31.1 [18.2 to 46.6]

5. Secondary Outcome: Percentage of Participants With Complete Remission With Partial Hematological Recovery (CRh*) During the First Two Treatment Cycles
Description: Participants were evaluated for efficacy at the end of each treatment cycle via a central bone marrow aspiration and local peripheral blood counts.
  Complete remission with partial hematological recovery (CRh*) was defined as meeting all 3 of the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease;
  * partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl.
  Participants without a post-baseline disease assessment were considered non-responders.
Time Frame: Approximately 12 weeks, as of the data cut-off date of 20 May 2015
Population: All participants who received an infusion of blinatumomab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
percentage of participants | 4.4 [0.5 to 15.1]

6. Secondary Outcome: Percentage of Participants With Complete Remission/Complete Remission With Partial Hematological Recovery/Complete Remission With Incomplete Hematological Recovery (CR/CRh*/CRi) During the First Two Treatment Cycles
Description: Efficacy was evaluated via a central bone marrow aspiration and local peripheral blood counts.
  Complete remission was defined as meeting the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease;
  * full recovery of peripheral blood counts: platelets > 100,000/μl, and absolute neutrophil count (ANC) > 1000/μl.
  Complete remission with partial hematological recovery was defined as meeting the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease;
  * partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl.
  Complete remission with incomplete hematologic recovery was defined as meeting all of the following criteria:
  * less than or equal to 5% blasts in the bone marrow;
  * no evidence of disease;
  * incomplete recovery of peripheral blood counts: platelets > 100,000/μl or ANC > 1000/μl.
  Participants without a post-baseline disease assessment were considered non-responders.
Time Frame: Approximately 12 weeks, as of the data cut-off date of 20 May 2015
Population: All participants who received an infusion of blinatumomab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
percentage of participants | 40.0 [25.7 to 55.7]

7. Secondary Outcome: Overall Survival
Description: Overall survival was assessed from the date the participant received the first infusion of blinatumomab until death from any cause or the date of the last follow-up.
  Participants still alive at the data cut-off date were censored on the last documented visit date or the date of the last contact when the patient was last known to have been alive.
Time Frame: From first dose of blinatumomab until the data cut-off date; median observation time was 8.8 months.
Population: All participants who received an infusion of blinatumomab
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
months | 7.1 [5.6 to NA] — Could not be estimated due to the low number of events at the time of analysis

8. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT) During Blinatumomab Induced Remission
Description: Participants who achieved remission (CR/CRh*) during the first 2 cycles of treatment and received an allogeneic HSCT.
Time Frame: Up to the data cut-of date of 20 May 2015; Maximum duration on study was 14.5 months.
Population: Participants who received an infusion of blinatumomab and had a CR/CRh* response during the first 2 cycles of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 16
percentage of participants | 43.8 [19.8 to 70.1]

9. Secondary Outcome: 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplant
Description: The analysis of 100-day mortality after allogeneic HSCT was assessed for participants who received an allogeneic HSCT while in remission (CR/CRh*) after 2 cycles of blinatumomab treatment and did not receive any additional antileukemic treatment. 100-day mortality after allogeneic HSCT was calculated relative to the date of allogeneic HSCT.
  The 100-day mortality rate after allogeneic HSCT was defined as the percentage of participants having died up to 100 days after allogeneic HSCT estimated using the estimated time to death in percent calculated by Kaplan-Meier methods. Participants alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive.
Time Frame: From the date of allogeneic HSCT until the data cut-off date of 20 May 2015; median observation time was 3.2 months.
Population: Participants who received allogeneic HSCT and were in remission with a CR/CRh* after 2 cycles of treatment and received the transplant without receiving any additional antileukemic medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 4
percentage of participants | 25.0 [3.9 to 87.2]

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity according to the CTCAE version 4.0, where Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE. Treatment-related adverse events (TRAEs) were those assessed by the investigator as possibly related to blinatumomab based on response to the question: Is there a reasonable possibility that the event may have been caused by blinatumomab or other protocol-specified therapies/procedures?
Time Frame: From the first dose of blinatumomab until 30 days after the last dose, up to the cut-off date of 20 May 2015; the median duration of treatment was 53.8 days.
Population: All participants who received an infusion of blinatumomab
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 45
participants
  Any adverse event | 45
  AE grade ≥ 3 | 37
  AE grade ≥ 4 | 18
  Serious adverse events | 28
  Leading to discontinuation of blinatumomab | 3
  Leading to interruption of blinatumomab | 16
  Fatal adverse events | 5
  Treatment-related adverse events | 41
  Treatment-related AE grade ≥ 3 | 20
  Treatment-related AE grade ≥ 4 | 7
  Treatment-related serious adverse events | 12
  TRAE leading to discontinuation of blinatumomab | 2
  TRAE leading to interruption of blinatumomab | 12
  Treatment-related fatal adverse events | 1

11. Secondary Outcome: Number of Participants Who Developed Anti-blinatumomab Antibodies
Description: Anti-blinatumomab binding antibodies were evaluated with a validated blinatumomab anti-drug antibody assay with the electrochemiluminescence detection technology.
Time Frame: Day 29 of each treatment period and 30 days after the last dose
Population: Participants with available post-baseline antibody results
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 29
participants | 0

12. Secondary Outcome: Steady State Concentration of Blinatumomab
Time Frame: Cycle 1, day 8, 6 to 8 hours after the dose step to 28 μg/day, and Cycle 2, day 1, 6 to 8 hours after blinatumomab infusion
Population: Participants with available serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 28
pg/mL
  Cycle 1 | 449 (125.6)
  Cycle 2 (n = 21) | 532 (128.7)

ADVERSE EVENTS:
Time Frame: From the first dose of blinatumomab until 30 days after the last dose, up to the cut-off date of 20 May 2015; the median duration of treatment was 53.8 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Blinatumomab
Serious Adverse Events (participants affected / at risk) | 28/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=45)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphoblastosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Aplasia (Congenital, familial and genetic disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Device infusion issue (General disorders) | 1
Device malfunction (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multi-organ failure (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Acute graft versus host disease (Immune system disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Catheter site infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 3
Lung infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=45)
Anaemia (Blood and lymphatic system disorders) | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 15
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Atrial fibrillation (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 9
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 6
Chest pain (General disorders) | 5
Chills (General disorders) | 4
Fatigue (General disorders) | 6
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 7
Pyrexia (General disorders) | 26
Cytokine release syndrome (Immune system disorders) | 3
Hypogammaglobulinaemia (Immune system disorders) | 3
Nasopharyngitis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Blood calcium decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 6
Confusional state (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.